CLINICAL TRIAL: NCT03253965
Title: The Effects of Auditory Cues on Gait Mechanics in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17-2089
Record Dates: First submitted 2017-08-11; First posted 2017-08-18 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking: Treadmill then Overground (Experimental): Walking while receiving auditory cueing intervals from a metronome and music. Testing performed using metronome normal, metronome slow, and metronome fast speed settings as well as music normal, music slow, and music fast tempos. Subjects will also walk with no auditory cueing.
  Interventions: Other: Metronome Normal; Other: Metronome Slow; Other: Metronome Fast; Other: Music Normal; Other: Music Slow; Other: Music Fast; Other: No Auditory cueing
- Walking: Overground, then Treadmill (Experimental): Walking while receiving auditory cueing intervals from a metronome and music. Testing performed using metronome normal, metronome slow, and metronome fast speed settings as well as music normal, music slow, and music fast tempos. Subjects will also walk with no auditory cueing.
  Interventions: Other: Metronome Normal; Other: Metronome Slow; Other: Metronome Fast; Other: Music Normal; Other: Music Slow; Other: Music Fast; Other: No Auditory cueing

INTERVENTIONS:
Other: Metronome Normal — Steps are timed with the beat of the metronome set to the subject's cadence
Other: Metronome Slow — Steps are timed with the beat of the metronome set to 85% of the subject's cadence
Other: Metronome Fast — Steps are timed with the beat of the metronome set to 115% of the subject's cadence
Other: Music Normal — Steps are timed with the beat of the music by a rhythm consistent with the subject's cadence
Other: Music Slow — Steps are timed with the beat of the music by a rhythm consistent with 85% of the subject's cadence
Other: Music Fast — Steps are timed with the beat of the music by a rhythm consistent with 115% of the subject's cadence
Other: No Auditory cueing — Steps are not timed with any auditory cue.

SUMMARY:
The purpose of this study is to determine how using auditory cues of a metronome and music at various frequencies impacts the gait mechanics in people with Parkinson's disease when walking over ground and on a treadmill.

The investigators will enroll a total of 40 participants: 30 subjects with a diagnosis of Parkinson's disease (10 in Stage 1, 10 in Stage 2, and 10 in Stage 3) and 10 unimpaired subjects.

Participants will complete 7 different treadmill walking conditions and overground walking conditions while the investigators measure step length, cadence, gait speed, and variability of movement.

ELIGIBILITY:
10 unimpaired controls and 30 subjects with Parkinson's Disease (described in detail below - see inclusion/exclusion criteria). The 30 subjects with Parkinson's Disease will be assigned into 3 groups (10 with H&Y Stage 1, 10 with H&Y Stage 2, and 10 with H&Y Stage 3).

Inclusion Criteria:

* Individuals with a diagnosis of Parkinson's Disease (made by movement disorders specialist) will be included in this study. Additional inclusion criteria include: self-reported ability to walk >10 m overground as well as walk on a treadmill for a total of 14 minutes with rest breaks as needed, and be classified as Stage 1, 2, or 3 on the Hoehn and Yahr Scale since these stages have the most independence with mobility (Goetz et. al, 2004).

Exclusion Criteria:

* Exclusion criteria include Hoehn and Yahr Stage 4 and 5, uncontrolled cardiorespiratory/metabolic disease (e.g., cardiac arrhythmia, uncontrolled hypertension or diabetes, orthostatic hypertension, chronic emphysema), or other neurological or orthopedic disorders that may affect walking. The investigators will also exclude participants with severe communication impairments, which could impede understanding of the purpose or procedures of the study or an inability to comply with experimental procedures.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Step Length | The entire duration of each condition, approximately 2 minutes each.
  The length of each step taken while walking on a treadmill or overground. It is the anteroposterior distance from one foot to the other at heel strike measured during walking under each condition.

SECONDARY OUTCOMES:
Cadence | The entire duration of each condition, approximately 2 minutes each.
  The number of steps taken per minute measured while walking on a treadmill or overground under each condition.
Gait speed | The entire duration of each condition, approximately 2 minutes each.
  The distance covered in a measured period of time (meters per second) while walking overground under each condition.
Movement variability | The entire duration of each condition, approximately 2 minutes each.
  The coefficient of variation of spatiotemporal measures (step timing and step length) while walking overground and on a treadmill under each condition.

CONTACTS AND LOCATIONS:
Overall Officials: Guneet Chawla, Principal Investigator — University of North Carolina, Chapel Hill; Michael Lewek, PT, PhD, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States